CLINICAL TRIAL: NCT06713187
Title: Role of Interleukin 23 in Systemic Lupus Erythematosus Related Interstial Lung Disease
Brief Title: Interleukin23 in Systemic Lupus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, khadiga Mahmoud Salem, resident doctor at clinical pathology department, Sohag University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh_Med__24_11_09MS
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Systemic Lupus Erythematosus Related Interstial Lung Disease
MeSH Terms: interventions — Interleukin-23

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 (Active Comparator): Patients with systemic lupus erythematosus without interstial lung disease.
  Interventions: Biological: interleukin 23
- group2 (Active Comparator): Patients with systemic lupus erythematosus with interstial lung disease.
  Interventions: Biological: interleukin 23
- group3 (Active Comparator): healthy control groups
  Interventions: Biological: interleukin 23

INTERVENTIONS:
Biological: interleukin 23 — assessment of interleukin 23 in Sera of patients using ELIZA

SUMMARY:
assement of interleukin 23 in serum of patients with systemic lupus erythematosus related interstial lung disease .

DETAILED DESCRIPTION:
for all patients detailed history taken clinical and rhumatological examination will be assessed and SLEDAI score will be collected from the case record of the patients&laboratory investigation included 1_erythrocytic sedimentation rate.2_complete blood count.3_interleukin23 .4_complement 3&4.5_Antinuclear Antibodies.6_Anti double stranded antibodies.7_full basic biochemical test(24 urine protien)8_high resolution computed tomography.

ELIGIBILITY:
Inclusion Criteria:

* patients with systemic lupus erythematous and patients with systemic lupus erythematosus with interstial lung disease.

Exclusion Criteria:

* patients with chest conditions rather than interstial lung disease &who receiving biological blocking antibodies& those treated with immunosuppressive drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
interleukin 23 | 2 years
  level of interleukin 23 in Sera of patients with systemic lupus erythematosus using ELIZA

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Sohag university hospital, Sohag
  - Sohag university, Sohag

REFERENCES:
- [Background] Yap DY, Lai KN. Cytokines and their roles in the pathogenesis of systemic lupus erythematosus: from basics to recent advances. J Biomed Biotechnol. 2010;2010:365083. doi: 10.1155/2010/365083. Epub 2010 May 6. PMID 20467470
- [Background] Haroon MM, Hegazy GA, Hassanien MA, Shaker O, Hussein WH. Significance of Interleukin 23 in Systemic Lupus Patients: Relation to Disease Activity and Damage Indices. Biologics. 2023 Jan 18;17:1-9. doi: 10.2147/BTT.S389021. eCollection 2023. PMID 36698375
- [Background] Sisto M, Lisi S. Interleukin-23 Involved in Fibrotic Autoimmune Diseases: New Discoveries. J Clin Med. 2023 Sep 1;12(17):5699. doi: 10.3390/jcm12175699. PMID 37685766
- [Background] Senoo S, Taniguchi A, Itano J, Oda N, Morichika D, Fujii U, Guo L, Sunami R, Kanehiro A, Tokioka F, Yoshimura A, Kiura K, Maeda Y, Miyahara N. Essential role of IL-23 in the development of acute exacerbation of pulmonary fibrosis. Am J Physiol Lung Cell Mol Physiol. 2021 Nov 1;321(5):L925-L940. doi: 10.1152/ajplung.00582.2020. Epub 2021 Sep 15. PMID 34524907